CLINICAL TRIAL: NCT00103363
Title: Lung Cancer Screening and Tissue Procurement
Brief Title: Sputum Cytology in Screening Heavy Smokers For Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Screening
Other Study IDs: 92-0392; UCHSC-92-392 (Other: University of Colorado Multiple Institutional Review Board)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cytology specimen collection procedure
Other: physiologic testing
Procedure: annual screening
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Screening tests, such as sputum cytology, may help doctors find tumor cells early and plan better treatment for lung cancer.

PURPOSE: This phase II trial is studying how well sputum cytology works in screening heavy smokers for lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Classify annual sputum samples cytologically in participants with or without airflow obstruction and a heavy smoking history.
* Correlate sputum cytological atypia (moderate atypia or worse) with lung cancer incidence in these participants.
* Correlate changes in sputum cytology (i.e., changes toward higher grades of atypia) with lung cancer incidence in these participants.

Secondary

* Determine other risk factors for lung cancer (e.g., diet, family history, smoking history, and medications) that may either confound or modify the association between sputum cytology and lung cancer risk in these participants.

OUTLINE: Two 3-day pooled sputum samples are collected for 6 consecutive days from participants by the spontaneous cough technique for cytopathological evaluation. Participants also complete a risk factor questionnaire and undergo a pulmonary function test by spirometry and a blood draw.

Participants complete a questionnaire updating smoking, vital, and lung cancer status and undergo sputum sample collection annually.

Participants are informed of sputum cytology results.

PROJECTED ACCRUAL: A total of 3,400 participants (2,900 with airflow obstruction and 500 without airflow obstruction) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current or ex-smoker with a lifetime history of cigarette smoking of ≥ 20 pack years, meeting 1 of the following criteria:

  * Airflow obstruction

    * FEV_1 < 75% predicted for age by spirometry
    * FEV_1/FVC ≤ 75% by spirometry
  * No airflow obstruction
* No history of lung cancer

PATIENT CHARACTERISTICS:

Age

* 25 and over

Performance status

* Not specified

Life expectancy

* More than 5 years

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No cancer within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3270 (Actual)
Dates: Start 1993-02; Primary Completion 1994-02 (Actual); Study Completion 1994-02 (Actual)

PRIMARY OUTCOMES:
Classification of annual sputum samples cytologically
Correlation of sputum cytological atypia (moderate atypia or worse) with lung cancer incidence
Correlation of changes in sputum cytology with lung cancer incidence

SECONDARY OUTCOMES:
Risk factors for lung cancer that may effect the association between sputum cytology and lung cancer risk

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kennedy, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center - Denver, Denver, Colorado, United States